CLINICAL TRIAL: NCT01660880
Title: Validation of Receptor Occupancy Simulation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jun Soo Kwon, Professor, Seoul National University Hospital
Other Study IDs: C-1205-094-410; A070001 (Other Grant/Funding Number: The Korean Healthcare Technology R&D Project)
Record Dates: First submitted 2012-07-23; First posted 2012-08-09 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Dopamine Receptor Occupancy; Medication Satisfaction; Prolactin Level; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- aripiprazole: Patient group who is treated with aripiprazole

SUMMARY:
* To estimate dopamine receptor occupancy by aripiprazole using computer simulation
* To measure dopamine receptor occupancy by aripiprazole in patients treated with the antipsychotics
* To validate the simulation result by comparing the receptor occupancy from the simulation with that from the patients

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of schizophrenia
* treated with aripiprazole or risperidone
* no change in dose of antipsychotics for at least 6 weeks
* total PANSS score should be below 80

Exclusion Criteria:

* Other psychiatric disorders rather than schizophrenia
* history of head trauma
* positive in urine hCG
* on antidepressant, anticholinergics or mood stabilizer

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with schizophrenia who is in the steady sate of antipsychotic treatment
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Dopamine receptor occupancy | 72 hrs after the last administration
  Measured using 11C-raclopride positron emission tomography

SECONDARY OUTCOMES:
Hamilton rating scale for depression | Baseline and 72 hours after the last administration
  HAM-D score
Barnes akathisia scale | Baseline and 72 hours after the last administration
  BAS score
Abnormal involuntary movement scale | Baseline and 72 hours after the last administration
  AIMS score
Simpson-Angus scale | Baseline and 72 hours after the last administration
  SAS score
Treatment satisfaction questionnaire for medication | Baseline and 72 hours after the last administration
  TSQM score
Medication satisfaction questionnaire | Baseline and 72 hours after the last administration
  MSQ score
N-back task | Baseline and 72 hours after the last administration
  To measure the change in working memory performance
Prolactin level | Baseline and 72 hours after the last administration
  To explore the effect of receptor occupancy on the blood prolactin level
Dopamine receptor occupancy | 3 hrs after the last administration
Dopamine receptor occupancy | 24 hrs after the last administration

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea